CLINICAL TRIAL: NCT01912326
Title: Prevention of Atrial Fibrillation by Optimized Overdrive Stimulation
Acronym: PAFOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B01- 408
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Bradycardia; Atrial Fibrillation
Keywords: pacemaker; atrial fibrillation
MeSH Terms: conditions — Bradycardia; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AF Suppression On (Active Comparator): AF Suppression Algorithm On, optimized AF Pacemaker Programming
  Interventions: Device: Pacemaker Implantation
- AF Suppression Off (Active Comparator): AF Suppression programmed Off, Optimized Pacemaker Programming
  Interventions: Device: Pacemaker Implantation

INTERVENTIONS:
Device: Pacemaker Implantation — Implantation of a dual chamber pacemaker
  Other Names: Pacemaker St. Jude Medical Identity DR Model 5370 or 5376

SUMMARY:
Evaluation of dynamic Atrial Overdrive Stimulation using the AF Suppression Algorithm to prevent atrial tachyarrhythmias in patients with more than 2% Auto Mode Switch Episodes with optimized pacemaker programming.

Hypothesis:

Dynamic atrial Overdrive (AF Suppression) reduces AT/AF Burden by 30% as compared to programming DDDR-(60) without AF Suppression when all other parameters are optimized.

DETAILED DESCRIPTION:
Atrial Fibrillation is the most common Heart Rhythm Disorder requiring therapy.

ELIGIBILITY:
Inclusion Criteria:

* indication for dual chamber pacemaker
* documented paroxysmal or persistent Atrial Fibrillation
* P-wave >1.0 mV in Sinus Rhythm or sufficient detection of AFib
* stable antyarrhythmic therapy
* age >= 19 years
* written informed consent
* implantation of a Identity DR 5370/5376 or later
* bipolar atrial lead

Exclusion Criteria:

* permanent AFib
* reversible etiology of AFib
* HYHA II or IV
* Coronary Artery disease with stable angina pectoris
* implanted ICD or planned implantation of a ICD
* cardiac surgery within the last 6 months or planned within 12 months
* live expectancy < 12 months
* pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2002-07; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Reduction of AT/AF Burden in the pacemaker diagnostics | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Bonn AdöR, Bonn, Germany